CLINICAL TRIAL: NCT05513638
Title: Safety and Accuracy of Artificial Intelligence-aided Precision MRI Assessment for the Optimization of Prostate Biopsy in Men With Suspicion of Prostate Cancer: a Multicenter Randomized Controlled Trial.
Brief Title: Artificial Intelligence-Based Computer-Aided Diagnosis of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-396
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: the Application of Artificial Intelligence in the Diagnosis of Prostate Cancer
Keywords: artificial intelligence; prostate cancer; magnetic resonance imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The First Affiliated Hospital of Nanjing Medical University
  Interventions: Diagnostic Test: the clinical use of artificial intelligence in the diagnosis of prostate cancer
- The First Affiliated Hospital of Soochow University
  Interventions: Diagnostic Test: the clinical use of artificial intelligence in the diagnosis of prostate cancer

INTERVENTIONS:
Diagnostic Test: the clinical use of artificial intelligence in the diagnosis of prostate cancer — Each study site will enroll consecutive eligible patients and randomize them to either (a) a group with human-based interpretation or (b) a group with human-artificial intelligence interactive interpretation, both of which are utilized as standards of care.

SUMMARY:
One-fifth of all men will develop clinically significant prostate cancers (CsPC) in their lifetime. An estimated 268,490 new prostate cancer (PCa) cases and 34,500 deaths are expected in the United States during the year 2022, making PCa the second most common cause of cancer-related deaths in men. MRI with the Prostate Imaging Reporting and Data System (PI-RADS) is a current widely used communicative tool for both CsPC detection and guiding targeted prostate biopsy. The high level of expertise required for accurate interpretation and persistent inter-reader variability has limited consistency and it has hindered the widespread adoption of PI-RADS. Artificial intelligence (AI) shows a broad prospect for medical interpretation and triage in various challenging tasks , including the PCa detection and staging with MRI. While rapid technical advances are furthering the application of AI medical imaging, their implementation in clinical practice remains a major hurdle. Besides, the prospect of data-derived AI tool is to assist human experts rather than replace them, and whether AI can match or exceed the human experts is still a matter of debate. Therefore, despite strong potential, there is urgent need for research to better quantify the accuracy, generalizability and clinical applicability before the clinical use of an AI in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicious of prostate cancer, presenting with an elevated prostatic specific antigen and/or abnormal digital rectal examination

Exclusion Criteria:

* (1) <60 years of age; (2) a previous surgery, radiotherapy or drug therapy for prostate cancer (interventions for benign prostatic hyperplasia or bladder outflow obstruction were deemed acceptable); (3) incomplete mp-MRI examination or artifacts of the images.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 60 years of age who are clinical suspicious of prostate cancer, presenting with an elevated prostatic specific antigen and/or abnormal digital rectal examination during the study enrollment period, will be eligible for inclusion. Patients will be excluded from screening if they are: (1) <60 years of age; (2) a previous surgery, radiotherapy or drug therapy for prostate cancer (interventions for benign prostatic hyperplasia or bladder outflow obstruction were deemed acceptable); (3) incomplete mp-MRI examination or artifacts of the images.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
biopsy or surgery confirmed newly-diagnosed prostate cancer and clinically significant prostate cancer | Aug,22nd,2022-Aug,22nd,2024
  Biopsy or surgery confirmed newly-diagnosed prostate cancer and clinically significant prostate cancer will serve as our primary outcome. Details of follow up and disease progression for a period of two years following mp-MRI will also be collected. For patients with no suspicious lesions on mp-MRI or biopsy-negative, follow-up prostatic specific antigen for a period of two years will also be collected.

SECONDARY OUTCOMES:
surgery confirmed T and N staging of prostate cancer | Aug,22nd,2022-Aug,22nd,2024
  surgery confirmed T and N staging of prostate cancer
positive rate of prostate biopsy | Aug,22nd,2022-Aug,22nd,2024
  positive rate of prostate biopsy in each arm
the total reviewing time | Aug,22nd,2022-Aug,22nd,2024
  The total reviewing time of radiologists will be measured in this aim. The reviewing time will be defined as the time from initiation of interpretating prostate mp-MRI to the time the radiologists finish reviewing and assigning a PI-RADS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Dong Zhang, Nanjing, China